CLINICAL TRIAL: NCT02214342
Title: Virtual Reality Based Balance Training in People With Mild Cognitive Impairment: A Pilot Study
Brief Title: Virtual Reality Based Balance Training in People With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Banner Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1401199972
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Distorted; Balance; Motor Deficit; Cognitive Deficit
MeSH Terms: conditions — Neurologic Manifestations; Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance Training (Experimental): Balance training will be conducted individually two times per week for 4 weeks. Each training session will include virtual reality tasks such as "ankle reaching" and "obstacle crossing" using a virtual obstacle shown on a computer screen. Each session will last 30 - 45 minutes.
  Interventions: Other: Balance Training
- Control (No Intervention): The control group will keep their normal activity without receiving any intervention.

INTERVENTIONS:
Other: Balance Training — Experimental: Balance Training Balance training will be conducted individually two times per week for 4 weeks. Each training session will include virtual reality tasks such as "ankle reaching" and "obstacle crossing" using a virtual obstacle shown on a computer screen. Each session will last 30 - 45 minutes.
  Arms: Balance Training

SUMMARY:
The aim of the present study is to evaluate an innovative virtual reality-based balance training intervention for improving clinically relevant motor performances (balance and gait) in people with mild cognitive impairment.

The investigators hypothesize that the virtual reality-based balance training intervention will improve balance and gait performances in people with mild cognitive impairment compared to a control group receiving usual care only.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Mild Cognitive Impairment
* willingness to provide informed consent

Exclusion Criteria:

* severe neurologic, cardiovascular, metabolic, or psychiatric disorders
* severe visual impairment
* severe cognitive impairment
* dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Postural Balance | 4 weeks
  Postural Balance during quiet standing for 30 seconds will be assessed using validated wearable sensor technology (BalanSens™)

SECONDARY OUTCOMES:
Gait performance | 4 weeks
  Gait performance will be measured using validated wearable sensor technology (LEGSys™)
Cognitive status | 4 weeks
  Changes in cognitive status will be measured by the Trail Making Test
Fear of falling | 4 weeks
  Fear of falling will be measured by the Falls Efficacy scale international (short form)
User experience | 4 weeks
  User experience will be measured using a standardized questionaire
Depressive signs | 4 weeks
  Depressive signs will be measured using the Center for Epidemiologic Studies Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Najafi, PhD, Principal Investigator — University of Arizona
Locations (1):
- Banner Sun Health Research Institute, Sun City, Arizona, United States